CLINICAL TRIAL: NCT02918357
Title: Gallium-68 PSMA-11 PET in Patients With Biochemical Recurrence
Acronym: PSMA BCR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Thomas Hope, Assistant Professor of Radiology and Biomedical Imaging, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 165510; NCI-2018-00039 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ga-68 labeled PSMA-11 PET (Experimental): PSMA PET imaging: Patients will receive Ga-68 labeled PSMA-11 PET and then undergo PET/CT or PET/MRI approximately 55-70 minutes later.
  Interventions: Drug: Ga-68 labeled PSMA-11 PET

INTERVENTIONS:
Drug: Ga-68 labeled PSMA-11 PET — Patients will be imaged using Ga-68 labeled PSMA-11 PET to determine if the presence of metastatic disease. Prostate Specific Membrane Antigen (PSMA) is a protein expressed on prostate cancer cells that can be imaged using small molecules that target this protocol.
  Other Names: Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled Glu-NH-CO-NH- Lys(Ahx)-HBED-CC; Ga-68 labeled Glu-urea- Lys(Ahx)-HBED-CC; Ga-68 labeled HBED-CC PSMA

SUMMARY:
The investigators are imaging patients with prostate cancer using a new PET imaging agent (Ga-68-PSMA-11) in order to evaluate it's ability to detection prostate cancer in patients with biochemical recurrence after prostatectomy and radiation therapy.

DETAILED DESCRIPTION:
Imaging and staging of prostate cancer is critical for surgical and treatment planning. Patients with suspected metastatic prostate cancer will be imaged using Gallium-68 labeled PSMA-11 in order to demonstrate its utility. The investigators plan to utilize this data to obtain further approvals of the Ga-68-PSMA-11 compound, so that this agent will become available for clinical imaging in prostate cancer patients. In the biochemical recurrence population, the primary objective is to determine the sensitivity and positive predictive value (PPV) on a per-patient and per-region-basis of 68Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological proven prostate adenocarcinoma.
* Rising prostate-specific antigen (PSA) after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy).

  * Post radical prostatectomy (RP) - American Urological Association (AUA) recommendation

    * PSA greater than 0.2 ng/mL measured more than 6 weeks after RP and,
    * Confirmatory persistent PSA greater than 0.2 ng/mL
  * Post-radiation therapy -ASTRO-Phoenix consensus definition

    * Nadir + greater than or equal to 2 ng/mL rise in PSA
* Karnofsky performance status of greater than 50 (or Eastern Cooperative Oncology Group (ECOG) /World Health Organization (WHO) equivalent).
* Age > 18.
* Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

* Investigational therapy for prostate cancer.
* Unable to lie flat, still or tolerate a PET scan.
* Prior history of any other malignancy within the last 2 years, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and superficial bladder cancer.
* Contraindication to furosemide administration including prior allergy or adverse reaction to furosemide or sulfa drugs. (Note: This exclusion criteria can be removed if Furosemide is omitted as part of the PET imaging protocol if a second-generation scatter correction is available for the used PET device).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ga-68 Labeled PSMA-11 Positron Emission Tomography (PET): Prostate Specific Membrane Antigen (PSMA) Positron Emission Tomography (PET) imaging: Patients will receive Ga-68 labeled PSMA-11 PET and then undergo PET/CT or PET/MRI approximately 55-70 minutes later.
  Ga-68 labeled PSMA-11 PET: Patients will be imaged using Ga-68 labeled PSMA-11 PET to determine if the presence of metastatic disease. Prostate Specific Membrane Antigen (PSMA) is a protein expressed on prostate cancer cells that can be imaged using small molecules that target this protocol.
Period: Overall Study
Arm/Group | Ga-68 Labeled PSMA-11 Positron Emission Tomography (PET)
Started | 385
Investigational Drug Administration | 385
PET/CT Scan | 385
Completed | 385
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 385
Age, Customized [Median (Full Range); unit: years]
  Age | 70 [45 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 385
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 318
  Black or African American | 8
  Native American and Alaska Native | 1
  Asian | 15
  Native Hawaiian | 0
  Other Pacific Islander | 0
  Other | 14
  Unknown | 29
Region of Enrollment [Number; unit: participants]
  United States | 385
Initial therapy [Count of Participants; unit: Participants]
  Prostatectomy only | 132
  Radiotherapy only | 124
  Prostatectomy and Salvage Radiotherapy | 129

OUTCOME MEASURES:

1. Primary Outcome: Positive Predictive Value (PPV) on a Per-patient Basis With Histologic Validation
Description: PPVs were calculated across the group on a per-patient basis on 68Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy and reported along with the corresponding two-sided 95% confidence intervals (CI). The CIs were constructed using the Wilson score method.
Time Frame: 1 month
Population: All subjects who received a 68Ga-PSMA-11 injection, had their 68Ga-PSMA-11 scan independently and blindly interpreted on a per patient basis. Per patient analyses included an evaluation of positive or negative for presence of localized prostate cancer (PCa).
Measure: Number (95% Confidence Interval); unit: percentage of times value is true
Groups:
- Pet Positive (Per Patient): Evaluate the PPV on a per-patient basis of 68Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy
Arm/Group | Pet Positive (Per Patient)
Number analyzed (Participants) | 125
percentage of times value is true | 0.90 [0.84 to 0.94]

2. Primary Outcome: Positive Predictive Value (PPV) on a Per-region Basis With Histologic Validation
Description: PPVs were calculated across the group on a per-region-basis on 68Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy and reported along with the corresponding two-sided 95% CIs. The CIs were constructed using the Wilson score method.
Time Frame: 1 month
Population: All subjects who received a 68Ga-PSMA-11 injection, had their 68Ga-PSMA-11 scan independently and blindly interpreted on a per region basis. Per region analyses included an evaluation of positive or negative for presence of PCa. Regional analyses included prostate bed, pelvic nodes, extrapelvic non-bone, and bone.
Measure: Number (95% Confidence Interval); unit: percentage of times value is true
Groups:
- Pet Positive (Per Region): Evaluate the PPV on a per-patient basis of 68Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy
Arm/Group | Pet Positive (Per Region)
Number analyzed (Participants) | 120
percentage of times value is true | 0.91 [0.85 to 0.95]

3. Secondary Outcome: PPVs on a Per-patient of 68Ga-PSMA-11 PET With Conventional Imaging Follow-up
Description: PPVs on a per-patient basis of 68Ga-PSMA-11 PET for detection of tumor location confirmed by conventional imaging follow-up were calculated and reported along with the corresponding two-sided 95% CI.
Time Frame: 1 month
Population: One hundred and twenty-five patients had confirmed imaging at follow-up for this analysis
Measure: Number (95% Confidence Interval); unit: percentage of times value is true
Arm/Group | Pet Positive (Per Patient)
Number analyzed (Participants) | 125
percentage of times value is true | 0.81 [0.69 to 0.89]

4. Secondary Outcome: PPVs on a Per-region of 68Ga-PSMA-11 PET With Conventional Imaging Follow-up
Description: PPVs on a per-region-basis of 68Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy and conventional imaging follow-up were calculated and reported along with the corresponding two-sided 95% CI.
Time Frame: 1 month
Population: Two-hundred and forty-nine patients had confirmed regional imaging in follow up for this sample.
Measure: Number (95% Confidence Interval); unit: percentage of times value is true
Arm/Group | Pet Positive (Per Patient)
Number analyzed (Participants) | 249
percentage of times value is true | 0.92 [0.88 to 0.95]

5. Secondary Outcome: Sensitivity on a Per-patient Basis
Description: Sensitivity, on a per-patient basis of 68Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy was calculated. The 95% CI was calculated using the Wilson score method.
Time Frame: 1 month
Population: Seventy-nine patients had confirmed patient histopathology validation for this analysis
Measure: Number (95% Confidence Interval); unit: percentage of sensitivity
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 79
percentage of sensitivity | 0.92 [0.84 to 0.96]

6. Secondary Outcome: Sensitivity on a Per-region Basis
Description: Sensitivity, on a per-region basis of 68Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy was calculated. The 95% CI was calculated using the Wilson score method.
Time Frame: 1 month
Population: Eighty-four patients had confirmed histopathology region validation for this analysis
Measure: Number (95% Confidence Interval); unit: percentage of sensitivity
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 84
percentage of sensitivity | 0.90 [0.82 to 0.95]

7. Secondary Outcome: Detection Rates of 68Ga-PSMA-11 PET Stratified by Prostate-specific Antigen (PSA) Value
Description: Detection rate was defined as proportion of 68Ga-PSMA-11 PET positive patients, independent of the reference standard stratified by PSA value (0.2-<0.5; 0.5-<1.0; 1.0-<2.0; 2.0-<5.0, and ≥5.0).
Time Frame: 1 month
Population: Portion of patients with 68Ga-PSMA-11 PET positive findings were stratified by PSA range and disease location in accordance with Prostate Magnetic Resonance Imaging Study (PROMIS)
Measure: Number; unit: percentage detected
Groups:
- PSA <0.5: Patients whom have a PSA nadir value of <0.5
- PSA 0.5 - <1.0: Patients whom have a PSA nadir value of 0.5 to <1.0
- PSA 1.0 - <2.0: Patients whom have a PSA nadir value of 1.0 to <2.0
- PSA 2.0 - <5.0: Patients whom have a PSA nadir value of 2.0 - <5.0
- PSA ≥5.0: Patients whom have a PSA nadir value of ≥5.0
Arm/Group | PSA <0.5 | PSA 0.5 - <1.0 | PSA 1.0 - <2.0 | PSA 2.0 - <5.0 | PSA ≥5.0
Number analyzed (Participants) | 82 | 41 | 53 | 103 | 106
percentage detected | 40 | 51 | 87 | 83 | 96

8. Secondary Outcome: Inter-reader Agreement Per-region
Description: Inter-reader reproducibility for positivity at region level was reported using the Fleiss' Kappa test for multiple readers. Kappa value varies from 0 (no agreement) to 1 (perfect agreement).
Time Frame: 1 month
Population: Patients included in the analyses were scanned to include all regions under review
Measure: Number (95% Confidence Interval); unit: kappa
Groups:
- Prostate Bed: Patients who have the prostate bed included in their study scan
- Pelvic Nodes: Patients who have the pelvic nodes included in their study scan
- Extrapelvic Soft Tissue: Patients who have the extrapelvic soft tissue included in their study scan
- Bone: Patients who have the pelvic bone included in their study scan
Arm/Group | Prostate Bed | Pelvic Nodes | Extrapelvic Soft Tissue | Bone
Number analyzed (Participants) | 385 | 385 | 385 | 385
kappa | 0.65 [0.61 to 0.70] | 0.73 [0.69 to 0.78] | 0.70 [0.65 to 0.74] | 0.78 [0.73 to 0.82]

9. Secondary Outcome: Percentage of Participants With Change in Clinical Management
Description: Clinical management changes were assessed using surveys of Intended Management to determine the percent change in clinical management after 68Ga-PSMA-11 PET.
Time Frame: Up to 1 year
Measure: Number; unit: Percentage of participants
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 382
Percentage of participants | 72

10. Secondary Outcome: Safety Assessment - Heart Rate
Description: Patient vital signs were measured before and after 68Ga-PSMA-11 injections and absolute mean change was calculated.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Pre-Infusion Heart Rate: All patients were assessed for safety measures that included Heart Rate before infusion
- Post-Infusion Heart Rate: All patients were assessed for safety measures that included Heart Rate after infusion
- Absolute Change in Heart Rate: All subjects had the absolute mean in heart rate calculated to assess for safety
Arm/Group | Pre-Infusion Heart Rate | Post-Infusion Heart Rate | Absolute Change in Heart Rate
Number analyzed (Participants) | 385 | 385 | 385
beats per minute | 67.8 (13.3) | 66.9 (13.6) | 0.9 (11.2)

11. Secondary Outcome: Safety Assessment - Blood Pressure
Description: Patient vital signs were measured before and after 68Ga-PSMA-11 injections and absolute mean change was calculated.
Time Frame: 1 day
Population: Pressure exerted by a 1 millimeter vertical column of mercury (Hg) at 0 degree Celsius is defined as (mmHg)
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Pre-Injection: All patients were assessed for safety measures that included blood pressure before infusion
- Post-Injection: All patients were assessed for safety measures that included blood pressure after infusion
- Absolute Mean Change: All subjects had the absolute mean in blood pressure calculated to assess for safety
Arm/Group | Pre-Injection | Post-Injection | Absolute Mean Change
Number analyzed (Participants) | 385 | 385 | 385
mmHg
  Systolic blood pressure | 137.8 (17.7) | 137.0 (17.4) | 1.0 (18.6)
  Diastolic blood pressure | 80.3 (33.8) | 81.1 (10.6) | 0.6 (34.0)

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events during and for 2 hours after radiotracer administration. Patients were also contacted by phone to assess for the development of delayed adverse events up to 24 hours after radiotracer administration.
Arm/Group | Ga-68 Labeled PSMA-11 PET
All-Cause Mortality (participants affected / at risk) | 0/385
Serious Adverse Events (participants affected / at risk) | 0/385
Other Adverse Events (participants affected / at risk) | 0/385

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-08-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT02918357/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT02918357/ICF_001.pdf